CLINICAL TRIAL: NCT05339867
Title: Prevent Maternal Mortality Using Mobile Technology (PM3)
Brief Title: Prevent Maternal Mortality Using Mobile Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Natalie Hernandez, Assistant Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00003016
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Post-Partum
Keywords: Postpartum Black mothers

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only the participants will be blinded to their assigned group. Immediately after participants have completed their baseline assessment, study staff will open a sealed envelope to identify the participants' group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers following Standard of Care (No Intervention): Participants randomized to this group will receive standard of Care for Postpartum. The standard of care control condition will be what women would typically get at hospital discharge (typically an Electronic Medical Record (EMR) generated document; a non-standardized, generalized brief review of how to care for self and the baby).
- Mother Using PM3 Intervention (Experimental): Participants in this group will be using the PM3 intervention. PM3 is a maternal mortality prevention and optimal reproductive health promotion mobile app created based on formative work with Black women to ultimately increase postpartum comorbidity self-management, promote timely provider notification of postpartum-related complications, and ensure access to social support and community resources.
  Interventions: Behavioral: Prevent Maternal Mortality using Mobile technology (PM3)

INTERVENTIONS:
Behavioral: Prevent Maternal Mortality using Mobile technology (PM3) — PM3: The app will include:
  1. integrated self-management and tailored health messaging feature
  2. support center based on social support gaps which will also provide a centralized place for identifying healthcare providers and facilities
  3. multimedia resource kit comprised of videos, current events, news feeds, podcasts, and support groups related to women's postpartum health and community resources
  4. a feature that will update women on maternal and reproductive health policies that impact women.
  Arms: Mother Using PM3 Intervention

SUMMARY:
Black women who reside in a rural area are at highest risk for maternal morbidity and mortality due to a combination of social and structural causes. The postpartum period is the most critical yet most neglected phase for preventing suboptimal or fatal maternal health outcomes. The goal of this project is to use a mobile app to provide personalized support and improve the lives of women during the early postpartum period. The information the study team gathers will help educate women and all who support them about the need to seek postpartum care and the impact postpartum care can have on pregnancy-related complications. Participation in this research requires taking part in a focus group discussion which will allow participants to share or the person that supports the participant's story and experience with postpartum complications and willingness to use and desired features of a postpartum mobile app.

DETAILED DESCRIPTION:
Black women in Georgia have the highest risk for adverse maternal outcomes, with a staggering 66.6 deaths per 100,000 live births, compared to 18.1 for Hispanic women and 43.2 for white women. In rural Georgia, these statistics are more profound, with Black women experiencing 126.7 deaths per 100,000 live births compared to 78.3 deaths for White women. These disparities have existed for centuries and have also widened significantly over the last several decades.

The proposed research aims to increase the effectiveness of postpartum discharge education and improve rural Black women's compliance with postpartum care recommendations by developing and testing a culturally-informed "mhealth intervention" entitled Prevent Maternal Mortality using Mobile technology (PM3).

ELIGIBILITY:
Inclusion Criteria:

* Participants self -identify as female
* Participants must self-identify as African American/Black
* Aged 18-45 years
* Can speak or read English
* Participants must be able to give consent.
* Own a smart phone
* Reside in or near Albany, LaGrange, or Waynesboro (within a 40 mile radius)
* Be in third trimester or recently had a baby (≤4 weeks postpartum)
* Can be contacted by phone or email after hospital discharge.

Exclusion Criteria:

* Women will be excluded if they have known unavailability to follow-up
* An active severe mental health condition, or developmental disability precluding informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of completion of postpartum healthcare visit ( Healthcare Resource utilization) | At weeks 4 to 6 postpartum
  Around 50% of the women receive a postpartum visit within that time. The study aims to increase postpartum visit attendance by 25% for a goal of 75%. The completion of a visit and other clinical outcomes will be confirmed by a medical chart review. This will be measured as number of participants completing the post partum healthcare visit.

SECONDARY OUTCOMES:
Changes in Current Life Situation | Baseline, month 3, month 6 and month 12
  All participants will complete a brief online socio-demographic survey containing closed-ended sociodemographic questions (e.g. marital status, educational attainment, employment status, health insurance status, total household income).
Changes in Women Sexual Health History | Baseline, month 3, month 6 and month 12
  All participants will complete a brief online socio-demographic survey containing closed-ended sociodemographic questions (e.g. marital status, educational attainment, employment status, health insurance status, total household income).
Changes in Blood pressure | Baseline, month 3, month 6 and month 12
  BP self-monitoring instructions will be provided when patients are enrolled, and patients will be expected to demonstrate understanding of how to take their own blood pressure and enter results into PM3. Using color-coded instructions, BP self-monitoring parameters will be used to create algorithms within the app. For instance, when patients input their BP, they will be prompted to retake the BP. If the second reading is outside the expected range, this will automatically trigger a request for a third reading (taken after 5 minutes). Persistent high or low readings will automatically trigger a message asking the participant to contact their obstetric provider or seek care at an emergency department. The app will provide notifications to remind patients to take their BP. Participants will be asked to take 1 BP measurement in the morning and 1 in the evening. Additionally, they will be asked to enter 1 weight measurement weekly.
Changes in Health related quality of life questionnaires (HRQoL) | Baseline, month 3, month 6 and month 12
  Health-related quality of life (HRQOL) is used to examine the impact of health status on quality of life. HRQOL is often measured by four core questions that asked about general health status and number of unhealthy days in the Behavioral Risk Factor Surveillance System (BRFSS) Unhealthy days are an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. The responses to questions 2 and 3 are combined to calculate a summary index of overall unhealthy days, with a logical maximum of 30 unhealthy days.
  Healthy days are the positive complementary form of unhealthy days. Healthy days estimates the number of recent days when a person's physical and mental health was good (or better) and is calculate by subtracting the number of unhealthy days from 30 days.
Changes in Hair cortisol levels | Baseline and 3 months
  Cortisol is a steroid hormone synthesized and secreted by the adrenal cortex and plays many important roles in regulating physiology including regulating the responses to acute and chronic stress. Hair is considered a reliable and stable measure of cortisol production and chronic stress. All study participants in the control and intervention arms will provide hair samples at baseline and at 3 months postpartum.
  During the study visit a strand of hair is cut, using fine scissors, as close to the participant's scalp as possible from a posterior vertex position. The hair is wrapped in aluminum foil to maintain the sample's integrity and avoid exposure to elements that might contaminate it. Hair samples are stored at room temperature in our lab space. On average, hair grows approximately one cm per month, allowing for approximately three months of aggregated cortisol data to be analyzed from each sample as a 3 cm hair segment reflects cumulative cortisol secretion over the past 3 months.
Edinburg Postpartum Depression Scale | Baseline, month 3, month 6 and month 12
  Early Depression Screening: 10-question Edinburg Postnatal Depression Scale (EPDS). This is a way of identifying patients at risk for perinatal depression. The EPDS is easy to administer and has proven to be an effective screening tool. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity. The EPDS score should not override clinical judgment. A careful clinical assessment should be carried out to confirm the diagnosis. The scale indicates how the mother has felt during the previous week. In doubtful cases it may be useful to repeat the tool after 2 weeks. The scale will not detect mothers with anxiety neuroses, phobias or personality disorders.
  QUESTIONS 1, 2, & 4 :Are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3.
  QUESTIONS 3, 5-10: Are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. Maximum score: 30 Possible Depression: 10 or greater
Changes in Promis-GSF | Baseline, month 3, month 6 and month 12
  Patient Reported Outcomes Measurement Information System (PROMIS) Global Short Form (GSF) instrument consists of ten global health items that represent five core PROMIS domains (physical function, pain, fatigue, emotional distress, social health). Four items are used to assess global physical health. Three of these are administered using five-category response scales, and one item (rating of pain on average) uses a response scale of 0-10 that is recoded to five categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5).
Discrimination & Stigma Scale | Baseline, month 3, month 6 and month 12
  The Discrimination and Stigma Scale (DISC) is measure of discrimination experienced based on having a mental health problem. The DISC has a 4-point Likert scale (not at all; a little; moderately; a lot) and assesses experiences of discrimination across 21 life domains including family, friends, dating or intimate relationships, housing and employment.
System Usability Scale | Baseline, month 3, month 6 and month 12
  The System Usability Scale (SUS) provides a quick, reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
  The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
  A SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret your results involves "normalizing" the scores to produce a percentile ranking.
Race-related stress (Index of Race-Related Stress-Brief)(IRRS-B) | Baseline, month 3, month 6 and month 12
  The 22-item IRRS-B aims to measure psychological stress related to experiences of racism for Black Americans in 3 subscales. The Cultural Racism subscale assesses the experience of racism when one's culture is vilified. The Institutional Racism subscale measures racism that is deeply entrenched in a particular institution's structure, policies, and processes. The Individual Racism subscale measures interpersonal racism. Participants will be asked to indicate their experience with and reaction to the events depicted in each item using a 5-point Likert-type scale (0 = this never happened to me; 1 = this event happened, but did not bother me; 2 = this event happened and I was slightly upset; 3 = this event happened and I was upset; 4 = this event happened and I was extremely upset). Items from each of the three subscales are summed to yield subscale scores, and higher scores indicate respondents endorsing a greater degree of stress as a result of their encounters with racism.
Changes in Sleep (Karolinska Sleep Questionnaire - KSS) | Baseline, month 3, month 6 and month 12
  This scale measures the subjective level of sleepiness at a particular time during the day. On this scale subjects indicate which level best reflects the psycho-physical sate experienced in the last 10 min. The KSS is a measure of situational sleepiness. It is sensitive to fluctuations. This is a 9-point scale (1 = extremely alert, 3= alert, 5 = neither alert nor sleepy, 7 = sleepy - but no difficulty remaining awake, and 9 = extremely sleepy - fighting sleep). Scores on the KSS increase with longer periods of wakefulness and it strongly correlate with the time of the day.
Medical Mistrust Index (MMI) | Baseline, month 3, month 6 and month 12
  The MMI includes 16 items on a 4-response Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree) (eg, "The US health care system has done harmful experiments on patients without their knowledge," "I trust that health care organizations keep up with the latest medical information"). Responses will be coded so that higher scores indicated higher mistrust.
Stressful Events Questionnaire | Baseline, month 3, month 6 and month 12
  The Stressful Life Events Screening Questionnaire (SLESQ) is a 13-item self-report measure for non-treatment seeking samples that assesses lifetime exposure to traumatic events. Eleven specific and two general categories of events, such as a life-threatening accident, physical and sexual abuse, witness to another person being killed or assaulted, are examined. For each event, respondents are asked to indicate whether the event occurred ("yes" or "no"), their age at time of the event, as well as other specific items related to the event, such as the frequency, duration, whether anyone died, or was hospitalization, etc.
Adverse Childhood Experiences (ACEs) questionnaire | Baseline, month 3, month 6 and month 12
  If the ACE score is 1-3 without ACE-Associated Health Conditions, the patient is at "intermediate risk" for toxic stress. If the ACE score is 1-3 and the patient has at least one ACE-associated condition, or if the ACE score is 4 or higher, the patient is at "high risk" for toxic stress.
General Perceived Self-Efficacy Scale | Baseline, month 3, month 6 and month 12
  The General Perceived Self-Efficacy Scale (GSES) is a ten-item scale that assessed the strength of an individual's belief in his/her own ability to respond to novel or difficult situations and to deal with any associated obstacles or setbacks. It is a self administered scale that normally takes 2-3 minutes to complete. For each item there is a four choice response from "not at all true" which scores 1, to "Exactly true" which scores 4. The scores of each item are summed to give a total score. The score on this scale reflects the strength of an individual's generalized efficacy belief. Thus the higher the score, the greater in the individual's generalized self-efficacy.
Social Support- The Medical Outcomes Study | Baseline, month 3, month 6 and month 12
  This brief, self-administered Social Support Survey instrument was developed for patients in the Medical Outcomes Study (MOS).The survey consists of four separate social support subscales and an overall functional social support index. A higher score for an individual scale or for the overall support index indicates more support.
  To obtain a score for each subscale, calculate the average of the scores for each item in the subscale.
  To obtain an overall support index, calculate the average of (1) the scores for all 18 items included in the four subscales, and (2) the score for the one additional item (see last item in the survey).
  To compare to published means in the article referenced below, scale scores can be transformed to a 0-100 scale using the following formula:100 x ((observed score - minimum possible score) / (maximum possible score - minimum possible score))
The Neighborhood Questionnaire | Baseline, month 3, month 6 and month 12
  The Neighborhood Questionnaire is a 16-item measure that assesses a parent's satisfaction with the family's neighborhood. The questionnaire explores sociability in the neighborhood, the neighborhood's stability, the quality of public services, neighborhood safety, the incidence of violent crime, drug traffic in the neighborhood, the parent's involvement with neighbors, and the parent's participation in neighborhood organizations. One item has nine response choices. Items ask about satisfaction level, quality, duration, quantity, level of involvement, and frequency. Three items are yes/no questions.
  This measure has three subscales: the Neighborhood Safety Subscale (items 1, 6, 10, 11, and 12), the Neighborhood Social Involvement Subscale (items 3, 4, 5, and 13), and the Public Services Subscale (items 8 and 9).
Appraisal of self-care agency Scale-Revised (ASAS-R) | Baseline, month 3, month 6 and month 12
  The Appraisal of Self-care Agency Scale (ASA-R) is one of the main instrument to assess self-care capacity. The ASA is a 24-item scale and each item is responded to on a five-point Likert type scale ranging from 1 (totally disagree) to 5 (totally agree) and with a total score that ranges from 24 to 120. The higher the score, the better the self-care agency.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Hernandez, PhD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University, Nell Hodgson Woodruff School of Nursing, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No